CLINICAL TRIAL: NCT05150119
Title: Correlation Between Altered Glycometabolic Status and Joint Inflammation in Diabetic Patients With Osteoarthritis Undergoing Knee Arthroplasty
Acronym: GLICO PG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: GLICO PG
Record Dates: First submitted 2021-11-27; First posted 2021-12-08 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: To Evaluate a Linear Positive Correlation Between Plasma HbA1c and Synovial IL-6 in Diabetic Patients

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Evaluation of Synovial IL-6 in diabetic patients with gonarthrosis — To evaluate if there is a linear positive correlation between plasma glycated hemoglobin concentration HbA1c and synovial IL-6 in diabetic patients
  Other Names: Evaluation of plasmatic HbA1c in diabetic patients with gonarthrosis

SUMMARY:
Evaluate the correlation between altered glycometabolic status and joint inflammation in diabetic patients with osteoarthritis undergoing knee replacement surgery

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients
* Patients with osteoarthritis awaiting knee replacement surgery
* Patients awaiting knee replacement surgery
* Patients who agree to sign informed consent

Exclusion Criteria:

* Patients less than 55 years of age.
* Patients over 85 years of age.
* Patients who are unable to understand and want.
* Patients with severe neurological disorders or with severe disabilities.
* Rheumatoid arthritis patients
* Cancer patients
* Patients suffering from chronic inflammatory bowel syndromes (RCU and Crohn's disease)
* Patients on immunosuppressive therapy

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population is made up of diabetic patients, of age, undergoing knee replacement surgery for osteoarthritis
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-11-15 (Actual); Primary Completion 2021-11-27 (Actual); Study Completion 2024-11-15 (Estimated)

PRIMARY OUTCOMES:
To evaluate if there is a linear positive correlation between plasma glycated hemoglobin concentration HbA1c and synovial IL-6 in diabetic patient | 2 day
  To evaluate if there is a linear positive correlation between plasma glycated hemoglobin concentration HbA1c and synovial IL-6 in diabetic patient

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Ortopedico Galeazzi, Milan, Italy